CLINICAL TRIAL: NCT04102020
Title: Multicenter, Phase 3 Study of Venetoclax and Azacitidine as Maintenance Therapy for Patients With Acute Myeloid Leukemia in First Remission After Conventional Chemotherapy
Brief Title: A Study of Oral Venetoclax Tablets and Oral Azacitidine as Maintenance Therapy in Adult Participants With Acute Myeloid Leukemia in First Remission After Conventional Chemotherapy
Acronym: VIALE-M
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: AbbVie (Industry)
Collaborators: Roche-Genentech (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M19-708; 2023-507221-42-00 (Other: EU CT)
Expanded Access: NCT03123029 (Available)
Record Dates: First submitted 2019-09-23; First posted 2019-09-25 (Actual); Results first posted 2025-08-20 (Actual); Last update posted 2025-08-20 (Actual); Status verified 2025-08

CONDITIONS: Acute Myeloid Leukemia (AML)
Keywords: Acute myeloid leukemia (AML); Venetoclax; Azacitidine (AZA); Maintenance Therapy; Conventional Chemotherapy; Best supportive care (BSC)
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — venetoclax; Azacitidine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- Part 1: Dose Confirmation (Experimental): Participants will receive venetoclax once daily (QD) (Days 1-28) for up to 24 cycles, azacitidine (AZA) QD on Days 1-5 of each 28 day cycle for up to 6 cycles.
  Interventions: Drug: Venetoclax; Drug: Azacitidine
- Part 3 (Dose Finding): Dose Escalation (Experimental): Participants will receive venetoclax QD for up to 24 cycles, AZA QD on Days 1 to 14 of each 28-day cycle for up to 24 cycles to determine recommended phase 3 dose (RPTD).
  Interventions: Drug: Venetoclax; Drug: Azacitidine
- Part 3 (Dose Finding): Safety Expansion (Experimental): Participants will receive venetoclax QD for up to 24 cycles, AZA QD on Days 1 to 14 of each 28-day cycle for up to 24 cycles at the RPTD.
  Interventions: Drug: Venetoclax; Drug: Azacitidine

INTERVENTIONS:
Drug: Venetoclax — Tablet: Oral
  Other Names: ABT-199; GDC-0199; Venclexta
Drug: Azacitidine — Subcutaneous (SC) or intravenous (IV) injection
  Arms: Part 1: Dose Confirmation
Drug: Azacitidine — Oral Tablet
  Arms: Part 3 (Dose Finding): Dose Escalation; Part 3 (Dose Finding): Safety Expansion

SUMMARY:
This study will be conducted in two parts. Part 1 will be the Dose Confirmation portion to determine recommended Phase 3 dose (RPTD) of venetoclax in combination with azacitidine (AZA). Part 3 will be the Dose Finding portion to determine RPTD of venetoclax in combination with AZA. Part 2 and Part 3 Randomization of the study were removed.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of newly diagnosed acute myeloid leukemia (AML).
* Participant meets the following disease activity criteria:

  * Confirmation of AML by World Health Organization (WHO) criteria (2016) and have confirmed complete remission (CR) or complete remission with incomplete blood count recovery (CRi) following completion of intensive induction and consolidation chemotherapies.
  * Achieved first CR + CRi within 120 days of first dose of study drug or be no more than 75 days since last dose of intensive conventional (including both induction and consolidation) chemotherapies.
  * AML has intermediate or poor risk cytogenetics per National Comprehensive Cancer Network (NCCN) 2016 criteria.
* Eastern Cooperative Oncology Group (ECOG) performance status <= 2.
* Participant must have adequate hematologic, renal, and liver function laboratory values as described in the protocol.

Exclusion Criteria:

* History of acute promyelocytic leukemia (APL).
* History of active central nervous system involvement with acute myeloid leukemia (AML).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2020-03-26 (Actual); Primary Completion 2022-09-29 (Actual); Study Completion 2026-06 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (156):
- United States (27):
  - Mitchell Cancer Institute /ID# 216443, Mobile, Alabama
  - Compassionate Cancer Care Research Group - Fountain Valley /ID# 216156, Fountain Valley, California
  - University of California, Los Angeles /ID# 219149, Los Angeles, California
  - Colorado Blood Cancer Institute /ID# 214280, Denver, Colorado
  - St. Alphonsus Regional Medical /ID# 216424, Boise, Idaho
  - Duplicate_Rush University Medical Center /ID# 218815, Chicago, Illinois
  - University of Kentucky Markey Cancer Center /ID# 215048, Lexington, Kentucky
  - Duplicate_Norton Cancer Institute /ID# 216401, Louisville, Kentucky
  - Tulane Medical Center - New Orleans /ID# 218166, New Orleans, Louisiana
  - Duplicate_Ochsner Clinic Foundation-New Orleans /ID# 214583, New Orleans, Louisiana
  - Tufts Medical Center /ID# 216110, Boston, Massachusetts
  - Massachusetts General Hospital /ID# 217307, Boston, Massachusetts
  - Duplicate_UMass Chan Medical School /ID# 218163, Worcester, Massachusetts
  - Oncology Hematology Associates (OHA) - Springfield /ID# 216351, Springfield, Missouri
  - Saint Louis University Cancer Center /ID# 218164, St Louis, Missouri
  - The John Theurer Cancer /ID# 215191, Hackensack, New Jersey
  - Rutgers Cancer Institute of New Jersey /ID# 239708, New Brunswick, New Jersey
  - Weill Cornell Medical College /ID# 214847, New York, New York
  - Providence Portland Medical Ct /ID# 216231, Portland, Oregon
  - Fox Chase Cancer Center /ID# 239372, Philadelphia, Pennsylvania
  - UPMC Hillman Cancer Ctr /ID# 214051, Pittsburgh, Pennsylvania
  - Duplicate_Prisma Health Cancer Institute-Faris Road /ID# 216066, Greenville, South Carolina
  - St Francis Cancer Center /ID# 216115, Greenville, South Carolina
  - Gibbs Cancer Center & Research /ID# 216192, Spartanburg, South Carolina
  - Tennessee Oncology-Nashville Centennial /ID# 218757, Nashville, Tennessee
  - Texas Oncology- Baylor Charles A. Sammons Cancer Center /ID# 214584, Dallas, Texas
  - University of Texas MD Anderson Cancer Center /ID# 225201, Houston, Texas
- Australia (11):
  - St George Hospital /ID# 215416, Kogarah, New South Wales
  - Liverpool Hospital /ID# 215415, Liverpool, New South Wales
  - Shoalhaven District Memorial Hospital /ID# 221973, Nowra, New South Wales
  - Wollongong Hospital /ID# 216071, Wollongong, New South Wales
  - Gold coast University Hospital /ID# 214650, Southport, Queensland
  - Toowoomba Hospital /ID# 217922, Toowoomba, Queensland
  - Princess Alexandra Hospital /ID# 238753, Woolloongabba, Queensland
  - Royal Adelaide Hospital /ID# 238754, Adelaide, South Australia
  - Box Hill Hospital /ID# 217622, Box Hill, Victoria
  - Barwon Health /ID# 217921, Geelong, Victoria
  - Perth Blood Institute Ltd /ID# 217531, Nedlands, Western Australia
- Canada (7):
  - Tom Baker Cancer Centre /ID# 214625, Calgary, Alberta
  - Duplicate_University of Alberta Hospital - Division of Hematology /ID# 215656, Edmonton, Alberta
  - Juravinski Cancer Centre /ID# 214623, Hamilton, Ontario
  - London Health Sciences Center- University Hospital /ID# 216055, London, Ontario
  - Ottawa Hospital Research Institute /ID# 214627, Ottawa, Ontario
  - University Health Network_Princess Margaret Cancer Centre /ID# 214624, Toronto, Ontario
  - Duplicate_McGill University Health Center Research Institute /ID# 215984, Montreal, Quebec
- China (13):
  - Beijing Friendship Hospital /ID# 216455, Beijing, Beijing Municipality
  - Chinese PLA General Hospital /ID# 216286, Beijing, Beijing Municipality
  - Peking University International Hospital /ID# 217439, Beijing, Beijing Municipality
  - Guangdong Provincial People's Hospital /ID# 216284, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University /ID# 215565, Guangzhou, Guangdong
  - Henan Cancer Hospital /ID# 215566, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technol /ID# 218046, Wuhan, Hubei
  - Tongji Hospital Tongji Medical College of HUST /ID# 216456, Wuhan, Hubei
  - Duplicate_Shanghai Tongji Hospital /ID# 218800, Shanghai, Shanghai Municipality
  - Tangdu Hospital of The Fourth Military Medical University, PLA /ID# 216283, Xi’an, Shanxi
  - West China Hospital, Sichuan University /ID# 216606, Chengdu, Sichuan
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sc /ID# 215558, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine /ID# 215564, Hangzhou, Zhejiang
- Czechia (3):
  - Fakultní Nemocnice Brno - Jihlavská /ID# 214807, Brno, Brno-mesto
  - Fakultni Nemocnice Ostrava /ID# 214809, Ostrava, Ostrava-mesto
  - Ustav hematologie a krevni transfuze /ID# 215137, Prague
- France (12):
  - Chu de Nice-Hopital L'Archet Ii /Id# 217368, Nice, Alpes-Maritimes
  - Duplicate_CHU Bordeaux - Hopital Haut Leveque /ID# 215150, Pessac, Gironde
  - CHRU Tours - Hopital Bretonneau /ID# 216186, Tours, Indre-et-Loire
  - CHRU Lille - Hopital Claude Huriez /ID# 217474, Lille, Nord
  - Duplicate_CHU de Nantes - Hotel Dieu /ID# 217367, Nantes, Pays de la Loire Region
  - Centre Hospitalier de la Cote Basque /ID# 216185, Bayonne, Pyrenees-Atlantiques
  - Centre Hospitalier du Mans /ID# 215148, Le Mans, Sarthe
  - Institut Gustave Roussy /ID# 215158, Villejuif, Val-de-Marne
  - Chu Angers /Id# 215151, Angers
  - Duplicate_Hopital Henri Mondor /ID# 215159, Créteil
  - Centre Hospitalier de Versailles André Mignot /ID# 215157, Le Chesnay
  - Hopital Avicenne - APHP /ID# 215152, Bobigny, Île-de-France Region
- Germany (5):
  - Universitaetsklinikum Giessen und Marburg /ID# 214734, Marburg, Hesse
  - Duplicate_Klinikum Chemnitz gGmbH /ID# 216073, Chemnitz, Saxony
  - Universitaetsklinikum Leipzig /ID# 214440, Leipzig, Saxony
  - Universitaetsklinikum Schleswig-Holstein Campus Luebeck /ID# 215173, Lübeck, Schleswig-Holstein
  - Universitaetsklinikum Halle (Saale) /ID# 221109, Halle
- Greece (6):
  - General Hospital of Athens Laiko /ID# 213869, Athens, Attica
  - University General Hospital Attikon /ID# 214298, Athens, Attica
  - University General Hospital of Heraklion PA.G.N.I /ID# 214075, Heraklion, Crete
  - General University Hospital of Alexandroupolis /ID# 213870, Alexandroupoli
  - General Hospital of Athens Evaggelismos and Ophthalmiatrio of Athens Polyclinic /ID# 213872, Athens
  - University General Hospital of Patras /ID# 213871, RION Patras Achaia
- Hungary (5):
  - Debreceni Egyetem-Klinikai Kozpont /ID# 214422, Debrecen, Hajdú-Bihar
  - Somogy Varmegyei Kaposi Mor Oktato Korhaz /ID# 214426, Kaposvár, Somogy County
  - Szabolcs-Szatmar-Bereg Varmegyei Oktatokorhaz /ID# 214425, Nyíregyháza, Szabolcs-Szatmár-Bereg
  - Vas Varmegyei Markusovszky Egyetemi Oktatokorhaz /ID# 215644, Szombathely, Vas County
  - Duplicate_Semmelweis Egyetem /ID# 214423, Budapest
- Israel (4):
  - Shaare Zedek Medical Center /ID# 239699, Jerusalem, Jerusalem
  - Hadassah Medical Center-Hebrew University /ID# 239700, Jerusalem, Jerusalem
  - Tel Aviv Sourasky Medical Center /ID# 239698, Tel Aviv, Tel Aviv
  - Rabin Medical Center /ID# 239696, Petah Tikva
- Italy (10):
  - Duplicate_IRCCS AOU di Bologna - Policlinico Sant'Orsola-Malpighi /ID# 213948, Bologna, Emilia-Romagna
  - Duplicate_Fondazione IRCCS Ca Granda Ospedale Maggiore Policlinico /ID# 214826, Milan, Milano
  - ASST Grande Ospedale Metropolitano Niguarda /ID# 213946, Milan, Milano
  - A.O.U. CITTA' DELLA SALUTE E DELLA SCIENZA DI TORINO - Ospedale Molinette /ID# 214505, Turin, Piedmont
  - Duplicate_Azienda Ospedaliero Universitaria Ospedali Riuniti di Ancona /ID# 213944, Ancona
  - ASST degli Spedali Civili di Brescia /ID# 214580, Brescia
  - Duplicate_A.O.U. Policlinico G. Rodolico S.Marco- Presidio G.Rodolico /ID# 214802, Catania
  - Duplicate_Azienda Ospedaliera di Rilievo Nazionale Antonio Cardarelli /ID# 213947, Napoli
  - Duplicate_Azienda Ospedaliera Universitaria Federico II /ID# 214278, Napoli
  - Ospedale S.Eugenio /ID# 214277, Rome
- Japan (15):
  - Japanese Red Cross Aichi Medical Center Nagoya Daiichi Hospital /ID# 215680, Nagoya, Aichi-ken
  - Aichi Cancer Center Hospital /ID# 215284, Nagoya, Aichi-ken
  - University of Fukui Hospital /ID# 215283, Yoshida-gun, Fukui
  - Duplicate_National Hospital Organization Kyushu Cancer Center /ID# 214841, Fukuoka, Fukuoka
  - Kyushu University Hospital /ID# 215286, Fukuoka, Fukuoka
  - Duplicate_Hokkaido University Hospital /ID# 215938, Sapporo, Hokkaido
  - Duplicate_National Hospital Organization Mito Medical Center /ID# 214699, Higashi Ibaraki-gun, Ibaraki
  - Tohoku University Hospital /ID# 214669, Sendai, Miyagi
  - Duplicate_Nagasaki University Hospital /ID# 214916, Nagasaki, Nagasaki
  - Duplicate_Okayama University Hospital /ID# 214840, Okayama, Okayama-ken
  - Osaka Metropolitan University Hospital /ID# 215225, Osaka, Osaka
  - Kindai University Hospital /ID# 214915, Osakasayama-shi, Osaka
  - Saitama Medical University International Medical Center /ID# 214823, Hidaka-shi, Saitama
  - NTT Medical Center Tokyo /ID# 214959, Shinagawa-ku, Tokyo
  - Yamagata University Hospital /ID# 214698, Yamagata, Yamagata
- Pan American Center for Oncology Trials, LLC /ID# 214953, Rio Piedras, Puerto Rico
- Russia (7):
  - Nizhny Novgorod Regional Clinical Hospital named N.A. Semashko /ID# 214309, Nizhny Novgorod, Nizhny Novgorod Oblast
  - Clinic of Immunopathology, SRIFCI /ID# 217937, Novosibirsk, Novosibirsk Oblast
  - Academician I.P. Pavlov First St. Petersburg State Medical University /ID# 215393, Saint Petersburg, Sankt-Peterburg
  - Regional Clinical Hospital of Yaroslavl /ID# 214318, Yaroslavl, Tatarstan, Respublika
  - P. Hertsen Moscow Oncology Research Institute /ID# 214312, Moscow
  - MMCC Kommunarka /ID# 215223, Moscow
  - Almazov National Medical Research Centre /ID# 214306, Saint Petersburg
- South Korea (4):
  - Duplicate_Pusan National University Hospital /ID# 213941, Busan, Busan Gwang Yeogsi
  - Seoul National University Bundang Hospital /ID# 215549, Seongnam-si, Gyeonggido
  - Seoul National University Hospital /ID# 213943, Seoul, Seoul Teugbyeolsi
  - Samsung Medical Center /ID# 213940, Seoul, Seoul Teugbyeolsi
- Spain (10):
  - Duplicate_Instituto Catalan de Oncologia (ICO) L'Hospitalet /ID# 214715, L'Hospitalet de Llobregat, Barcelona
  - Duplicate_Hospital Universitario de Navarra /ID# 214788, Pamplona, Navarre
  - Hospital Santa Creu i Sant Pau /ID# 214714, Barcelona
  - Duplicate_Hospital Universitario Reina Sofia /ID# 214786, Córdoba
  - Hospital Universitario Infanta Leonor /ID# 214843, Madrid
  - MD Anderson Madrid /ID# 214477, Madrid
  - Hospital Universitario Ramon y Cajal /ID# 214684, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz /ID# 214933, Madrid
  - Hospital Universitario 12 de Octubre /ID# 214789, Madrid
  - Hospital Universitario Virgen de la Victoria /ID# 214713, Málaga
- Taiwan (4):
  - National Taiwan University Hospital /ID# 213939, Taipei City, Taipei
  - Kaohsiung Medical University Chung-Ho Memorial Hospital /ID# 213953, Kaohsiung City
  - China Medical University Hospital /ID# 213952, Taichung
  - Linkou Chang Gung Memorial Hospital /ID# 213951, Taoyuan
- Turkey (Türkiye) (5):
  - Gulhane Askeri Tip Academy /ID# 214242, Ankara
  - Ankara Univ Medical Faculty /ID# 214239, Ankara
  - Istanbul Universitesi-Cerrahpasa Cerrahpasa Tip Fakultesi /ID# 215525, Istanbul
  - Erciyes University Medical Faculty /ID# 214240, Kayseri
  - Karadeniz University /ID# 214241, Trabzon
- United Kingdom (7):
  - Leicester Royal Infirmary /ID# 215924, Leicester, England
  - Disc_Barts Health NHS Trust - The Royal London Hospital /ID# 215909, London, Greater London
  - Duplicate_UCLH NHS Foundation Trust - University College Hospital /ID# 215921, London, Greater London
  - Dup_Guys and St Thomas NHS Foundation Trust - Guy's Hospital /ID# 215908, London, Greater London
  - Cardiff & Vale University Health Board /ID# 215906, Cardiff, Wales
  - University Hospitals Birmingham NHS Foundation Trust /ID# 215910, Birmingham
  - University Hospitals Bristol /ID# 215911, Bristol

IPD SHARING:
Plan to Share IPD: Yes
AbbVie is committed to responsible clinical trial data sharing. This includes access to anonymized, individual and trial-level data (analysis data sets), as well as other information.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: For details on when studies are available for sharing visit https://vivli.org/ourmember/abbvie/
Access Criteria: To learn more about the process, or to submit a request, visit the following link https://www.abbvieclinicaltrials.com/hcp/data-sharing/
URL: https://vivli.org/ourmember/abbvie/

REFERENCES:
- [Derived] Ivanov V, Yeh SP, Mayer J, Saini L, Unal A, Boyiadzis M, Hoffman DM, Kang K, Addo SN, Mendes WL, Fathi AT. Design of the VIALE-M phase III trial of venetoclax and oral azacitidine maintenance therapy in acute myeloid leukemia. Future Oncol. 2022 Aug;18(26):2879-2889. doi: 10.2217/fon-2022-0450. Epub 2022 Jul 19. PMID 35852098
- [Derived] Shallis RM, Podoltsev NA. Maintenance therapy for acute myeloid leukemia: sustaining the pursuit for sustained remission. Curr Opin Hematol. 2021 Mar 1;28(2):110-121. doi: 10.1097/MOH.0000000000000637. PMID 33394722
- See also: Related Info — https://www.abbvieclinicaltrials.com/study/?id=M19-708

RESULTS

PARTICIPANT FLOW:
Groups:
- Part 1: Venetoclax 400 mg + Azacitidine 20 mg/m^2; Part 1: Venetoclax 400 mg + Azacitidine 36 mg/m^2; Part 1: Venetoclax 400 mg + Azacitidine 50 mg/m^2: Participants will receive venetoclax once daily (QD) (Days 1-28) for up to 24 cycles, azacitidine (AZA) QD on Days 1-5 of each 28 day cycle for up to 6 cycles.
  Venetoclax: Tablet: Oral
  Azacitidine: Subcutaneous (SC) or intravenous (IV) injection
- Part 3: Dose Level 1 - Venetoclax 400mg + CC-486 200mg: Participants will receive venetoclax QD for up to 24 cycles, AZA QD on Days 1 to 14 of each 28-day cycle for up to 24 cycles to determine recommended phase 3 dose (RPTD).
  Venetoclax: Tablet: Oral
  Azacitidine: Oral Tablet
- Part 3: Dose Level 2 - Venetoclax 400mg + CC-486 300mg: Participants will receive venetoclax QD for up to 24 cycles, AZA QD on Days 1 to 14 of each 28-day cycle for up to 24 cycles at the RPTD.
  Venetoclax: Tablet: Oral
  Azacitidine: Oral Tablet
Period: Overall Study
Arm/Group | Part 1: Venetoclax 400 mg + Azacitidine 20 mg/m^2 | Part 1: Venetoclax 400 mg + Azacitidine 36 mg/m^2 | Part 1: Venetoclax 400 mg + Azacitidine 50 mg/m^2 | Part 3: Dose Level 1 - Venetoclax 400mg + CC-486 200mg | Part 3: Dose Level 2 - Venetoclax 400mg + CC-486 300mg
Started | 23 | 23 | 20 | 30 | 16
Completed (Data included are subject to a cutoff date of 05OCT2022.) | 0 | 0 | 0 | 0 | 0
Not Completed | 23 | 23 | 20 | 30 | 16
Not completed — Adverse Event | 1 | 0 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 0 | 1 | 1 | 1 | 1
Not completed — Death | 1 | 4 | 1 | 1 | 0
Not completed — Physician Decision | 1 | 2 | 2 | 0 | 1
Not completed — COVID-19 Infection | 1 | 0 | 0 | 0 | 0
Not completed — Not disclosed | 5 | 3 | 8 | 0 | 1
Not completed — MIssing | 1 | 0 | 1 | 1 | 1
Not completed — Continuing in ongoing study | 13 | 13 | 7 | 26 | 12

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Part 1: Venetoclax 400 mg + Azacitidine 20 mg/m^2 | Part 1: Venetoclax 400 mg + Azacitidine 36 mg/m^2 | Part 1: Venetoclax 400 mg + Azacitidine 50 mg/m^2 | Part 3: Dose Level 1 - Venetoclax 400mg + CC-486 200mg | Part 3: Dose Level 2 - Venetoclax 400mg + CC-486 300mg | Total
Number analyzed (Participants) | 23 | 23 | 20 | 30 | 16 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.1 (13.97) | 57.3 (13.89) | 55.6 (16.26) | 58.8 (12.70) | 54.1 (16.94) | 55.78 (14.75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 10 | 16 | 6 | 56
  Male | 10 | 12 | 10 | 14 | 10 | 56
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 6 | 6 | 8 | 5 | 2 | 27
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0 | 0
  White | 17 | 16 | 12 | 25 | 14 | 84
  More than one race | 0 | 1 | 0 | 0 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-Limiting Toxicities (DLTs) of Venetoclax in Combination With Azacitidine (AZA) (Part 1)
Description: DLTs are any of the hematologic, nonhematologic toxicities, adverse events (AEs) occurring following administration of venetoclax as described in the protocol and evaluated by the Investigator and the sponsor.
Time Frame: Up to 28 days (Cycle 1)
Population: Data included are subject to a cutoff date of 05Oct2022.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 1: Venetoclax 400 mg + Azacitidine 20 mg/m^2 | Part 1: Venetoclax 400 mg + Azacitidine 36 mg/m^2 | Part 1: Venetoclax 400 mg + Azacitidine 50 mg/m^2
Number analyzed (Participants) | 22 | 19 | 16
Participants
  Neutropenia | 3 | 4 | 4
  Leukopenia | 1 | 0 | 0
  Thrombocytopenia | 1 | 0 | 0
  Platelet count decreased | 1 | 0 | 0

2. Primary Outcome: Number of Participants With DLTs of Venetoclax in Combination With Oral AZA (Part 3 Dose Finding Portion)
Description: DLTs are hematologic toxicities consisting of any Grade ≥ 3 neutropenia or thrombocytopenia lasting more than 7 days and nonhematologic toxicities as described in the protocol and evaluated by the Investigator and the Sponsor. In addition, AEs that lead to omitting > 20% of the scheduled dose within the cycle is considered as a DLT unless clearly related to underlying disease. Treatment delay due to toxicity lasting greater than 14 days since the last dose of Venetoclax is also considered a DLT.
Time Frame: Up to 28 days (Cycle 1)
Population: Data included are subject to a cutoff date of 05Oct2022.
Measure: Count of Participants; unit: Participants
Arm/Group | Part 3: Dose Level 1 - Venetoclax 400mg + CC-486 200mg | Part 3: Dose Level 2 - Venetoclax 400mg + CC-486 300mg
Number analyzed (Participants) | 14 | 11
Participants
  Neutropenia | 1 | 2
  Thrombocytopenia | 1 | 1
  Febrile neutropenia | 0 | 1
  Fatigue | 0 | 1
  Neutrophil count decreased | 1 | 1
  Platelet count decreased | 0 | 1
  Dizziness | 1 | 0

ADVERSE EVENTS:
Time Frame: All-cause mortality and adverse event tables include events reported from the time of informed consent to the interim cutoff date of 05OCT2022. The median time on follow-up was 446, 687, 389 days for Part 1 VEN400_AZA20, VEN400_AZA36, VEN400_AZA50 and 67.5, 275 days for Part 3 Dose Level 1 (VEN400_CC200), Dose Level 2 (VEN400_CC300), respectively.
Arm/Group | Part 1: Venetoclax 400 mg + Azacitidine 20 mg/m^2 | Part 1: Venetoclax 400 mg + Azacitidine 36 mg/m^2 | Part 1: Venetoclax 400 mg + Azacitidine 50 mg/m^2 | Part 3: Dose Level 1 - Venetoclax 400mg + CC-486 200mg | Part 3: Dose Level 2 - Venetoclax 400mg + CC-486 300mg
All-Cause Mortality (participants affected / at risk) | 3/23 | 5/23 | 1/20 | 1/30 | 1/16
Serious Adverse Events (participants affected / at risk) | 5/23 | 7/23 | 5/20 | 5/30 | 3/16
Other Adverse Events (participants affected / at risk) | 21/23 | 22/23 | 20/20 | 29/30 | 16/16
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Venetoclax 400 mg + Azacitidine 20 mg/m^2 (N=23) | Part 1: Venetoclax 400 mg + Azacitidine 36 mg/m^2 (N=23) | Part 1: Venetoclax 400 mg + Azacitidine 50 mg/m^2 (N=20) | Part 3: Dose Level 1 - Venetoclax 400mg + CC-486 200mg (N=30) | Part 3: Dose Level 2 - Venetoclax 400mg + CC-486 300mg (N=16)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 1 (2) | 0 (0) | 0 (0) | 2 (3)
LEUKOPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 0 (0)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 2 (2) | 1 (1) | 1 (2) | 1 (1) | 0 (0)
ATRIAL FIBRILLATION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
CARDIAC TAMPONADE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COLITIS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ANORECTAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
BACILLUS INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
CELLULITIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 PNEUMONIA (Infections and infestations) | 1 (2) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
PSEUDOMONAL SEPSIS (Infections and infestations) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
EUGLYCAEMIC DIABETIC KETOACIDOSIS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
HAEMORRHAGIC STROKE (Nervous system disorders) | 1 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: Venetoclax 400 mg + Azacitidine 20 mg/m^2 (N=23) | Part 1: Venetoclax 400 mg + Azacitidine 36 mg/m^2 (N=23) | Part 1: Venetoclax 400 mg + Azacitidine 50 mg/m^2 (N=20) | Part 3: Dose Level 1 - Venetoclax 400mg + CC-486 200mg (N=30) | Part 3: Dose Level 2 - Venetoclax 400mg + CC-486 300mg (N=16)
ANAEMIA (Blood and lymphatic system disorders) | 4 (4) | 8 (19) | 7 (16) | 3 (3) | 4 (15)
FEBRILE NEUTROPENIA (Blood and lymphatic system disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
LEUKOPENIA (Blood and lymphatic system disorders) | 6 (23) | 7 (34) | 7 (34) | 4 (4) | 4 (11)
LYMPHOPENIA (Blood and lymphatic system disorders) | 1 (10) | 2 (3) | 4 (16) | 1 (1) | 0 (0)
NEUTROPENIA (Blood and lymphatic system disorders) | 13 (75) | 16 (69) | 16 (65) | 10 (23) | 9 (28)
THROMBOCYTOPENIA (Blood and lymphatic system disorders) | 8 (21) | 13 (38) | 11 (46) | 7 (14) | 6 (14)
TINNITUS (Ear and labyrinth disorders) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
VERTIGO (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 1 (1) | 1 (2) | 0 (0)
VISION BLURRED (Eye disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
ABDOMINAL PAIN (Gastrointestinal disorders) | 3 (4) | 1 (1) | 0 (0) | 2 (3) | 2 (6)
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 5 (7) | 0 (0) | 2 (3) | 4 (4) | 0 (0)
ANAL FISTULA (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
APHTHOUS ULCER (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
CONSTIPATION (Gastrointestinal disorders) | 1 (1) | 5 (5) | 1 (1) | 8 (10) | 3 (6)
DENTAL CARIES (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
DIARRHOEA (Gastrointestinal disorders) | 6 (14) | 2 (3) | 5 (5) | 13 (15) | 7 (23)
DYSPEPSIA (Gastrointestinal disorders) | 1 (1) | 3 (3) | 1 (1) | 1 (1) | 2 (2)
FLATULENCE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
FREQUENT BOWEL MOVEMENTS (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 0 (0) | 2 (2) | 1 (1) | 1 (1) | 0 (0)
GINGIVAL BLEEDING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GINGIVAL PAIN (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GINGIVAL SWELLING (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NAUSEA (Gastrointestinal disorders) | 6 (15) | 3 (3) | 4 (8) | 15 (20) | 9 (18)
TOOTHACHE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VOMITING (Gastrointestinal disorders) | 3 (5) | 2 (5) | 0 (0) | 9 (19) | 9 (14)
ASTHENIA (General disorders) | 0 (0) | 0 (0) | 1 (1) | 3 (5) | 2 (6)
CHEST PAIN (General disorders) | 0 (0) | 1 (1) | 1 (1) | 1 (1) | 0 (0)
FATIGUE (General disorders) | 2 (2) | 2 (2) | 1 (1) | 4 (4) | 4 (5)
INFLUENZA LIKE ILLNESS (General disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 3 (3)
INJECTION SITE REACTION (General disorders) | 0 (0) | 1 (1) | 1 (4) | 0 (0) | 0 (0)
MUCOSAL INFLAMMATION (General disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0) | 0 (0)
OEDEMA PERIPHERAL (General disorders) | 2 (3) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
PAIN (General disorders) | 1 (1) | 3 (5) | 1 (1) | 1 (1) | 1 (1)
PYREXIA (General disorders) | 2 (2) | 2 (2) | 3 (8) | 0 (0) | 0 (0)
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1) | 0 (0)
HYPERTRANSAMINASAEMIA (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
SEASONAL ALLERGY (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ASYMPTOMATIC COVID-19 (Infections and infestations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
BACTERIAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
BRONCHITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 2 (2) | 5 (5) | 2 (2) | 3 (3) | 6 (6)
CYSTITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GINGIVITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HERPES SIMPLEX (Infections and infestations) | 0 (0) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
HERPES ZOSTER (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
ORAL HERPES (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (1)
PERIORBITAL INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
PHARYNGITIS (Infections and infestations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PHARYNGOTONSILLITIS (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 2 (2) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
RHINITIS (Infections and infestations) | 0 (0) | 3 (3) | 1 (1) | 0 (0) | 0 (0)
SKIN INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
SOFT TISSUE INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
STAPHYLOCOCCAL SEPSIS (Infections and infestations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
TINEA INFECTION (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 (1) | 0 (0) | 2 (2) | 1 (1) | 2 (2)
URINARY TRACT INFECTION (Infections and infestations) | 3 (3) | 3 (3) | 0 (0) | 0 (0) | 1 (1)
LIMB INJURY (Injury, poisoning and procedural complications) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
PROCEDURAL PAIN (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (3) | 4 (14) | 2 (4) | 1 (1) | 2 (3)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 1 (1) | 3 (4) | 1 (1) | 0 (0) | 1 (2)
BILIRUBIN CONJUGATED INCREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (2)
BLOOD ALKALINE PHOSPHATASE INCREASED (Investigations) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (3)
BLOOD BILIRUBIN INCREASED (Investigations) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
BLOOD CREATININE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
BLOOD LACTATE DEHYDROGENASE INCREASED (Investigations) | 0 (0) | 1 (1) | 0 (0) | 2 (5) | 0 (0)
BLOOD UREA INCREASED (Investigations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NEUTROPHIL COUNT DECREASED (Investigations) | 3 (28) | 1 (1) | 4 (19) | 3 (19) | 4 (50)
PLATELET COUNT DECREASED (Investigations) | 4 (19) | 3 (7) | 3 (11) | 3 (7) | 5 (22)
WEIGHT DECREASED (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (3)
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 5 (33) | 1 (6) | 3 (12) | 1 (14) | 3 (6)
DECREASED APPETITE (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 1 (4)
DYSLIPIDAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
HYPERURICAEMIA (Metabolism and nutrition disorders) | 0 (0) | 2 (2) | 3 (6) | 0 (0) | 0 (0)
HYPOCALCAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HYPOKALAEMIA (Metabolism and nutrition disorders) | 2 (2) | 3 (6) | 2 (2) | 1 (1) | 0 (0)
HYPOMAGNESAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
HYPOURICAEMIA (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 3 (4) | 1 (2) | 3 (6) | 2 (2) | 0 (0)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1) | 2 (3) | 1 (1) | 1 (1) | 0 (0)
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 1 (1) | 3 (3) | 0 (0) | 0 (0) | 0 (0)
ACROCHORDON (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
DIZZINESS (Nervous system disorders) | 5 (5) | 1 (1) | 1 (1) | 3 (3) | 0 (0)
HEADACHE (Nervous system disorders) | 0 (0) | 4 (4) | 2 (2) | 4 (5) | 2 (2)
LETHARGY (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PARAESTHESIA (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2)
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
INSOMNIA (Psychiatric disorders) | 2 (2) | 2 (2) | 0 (0) | 0 (0) | 1 (1)
NEPHROLITHIASIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
BENIGN PROSTATIC HYPERPLASIA (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
VULVOVAGINAL DRYNESS (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
COUGH (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 3 (3) | 0 (0) | 1 (2)
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
EPISTAXIS (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (2) | 1 (1) | 0 (0) | 0 (0)
OROPHARYNGEAL PAIN (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PRODUCTIVE COUGH (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
RHINITIS ALLERGIC (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ASTEATOSIS (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
DERMAL CYST (Skin and subcutaneous tissue disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
ECZEMA (Skin and subcutaneous tissue disorders) | 1 (2) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
ERYTHEMA (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MACULE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PAPULE (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
PRURITUS (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (3) | 5 (5) | 1 (1) | 3 (4)
PURPURA (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 4 (5) | 0 (0) | 2 (3) | 1 (1) | 3 (3)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (5) | 0 (0) | 1 (1) | 0 (0)
SKIN EXFOLIATION (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HAEMATOMA (Vascular disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
HYPERTENSION (Vascular disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (4) | 0 (0)
SUPERFICIAL VEIN THROMBOSIS (Vascular disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2024-04-26): https://cdn.clinicaltrials.gov/large-docs/20/NCT04102020/Prot_000.pdf
  • Statistical Analysis Plan (2020-09-21): https://cdn.clinicaltrials.gov/large-docs/20/NCT04102020/SAP_001.pdf